CLINICAL TRIAL: NCT06530667
Title: A Prospective Clinic Study to Evaluate the Effectiveness Safety and Feasibility of the Broadband Collaborative Pulse Ablation Instrument in Treating Malignant Pulmonary Nodules
Brief Title: Broadband Collaborative Pulse Ablation Instrument Treating Malignant Pulmonary Nodules
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-IR-110R
Record Dates: First submitted 2024-07-22; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Lung Neoplasm Malignant; Secondary Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Patients treated by broadband collaborative pulse ablation
  Interventions: Device: broadband collaborative pulse ablation

INTERVENTIONS:
Device: broadband collaborative pulse ablation — Via CT guided, patients with malignant pulmonary nodules would be treated by broadband collaborative pulse ablation

SUMMARY:
Effectiveness safety and feasibility of the broadband collaborative pulse ablation instrument in treating malignant pulmonary nodules

DETAILED DESCRIPTION:
This clinical trial is to observe the safety and efficacy of the broadband synergistic pulse ablation device for treating malignant pulmonary nodules, and to provide reference data for the development of formal trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18 and 70 years old with no gender limitation;
2. Malignant pulmonary nodules diagnosed by cytology and/or histopathology, or the number of tumors ≤3. The pulmonary nodules were oligometastatic and the primary lesions were stable, with no uncontrolled metastasis to other sites;
3. Surgery is not available or the patient refuses surgical treatment;
4. Nodules' Maximum diameter≤2cm;
5. ECOG score≤2;
6. Patients understood the trial procedure and voluntarily signed informed consent.

Exclusion Criteria:

1. An electronic device is implanted near the target area or an implanted pacemaker or defibrillator is present in the body;
2. Coagulation dysfunction with severe bleeding tendency and short-term correction (prothrombin time >18s, prothrombin activity <40%, platelet <80×109 /L);
3. Patient who can not stop taking Antiplatelet and anticoagulant drugs 5 days before surgery;
4. Severe pulmonary fibrosis and pulmonary hypertension;
5. Patients with poor control of pleural effusion;
6. Patients with serious insufficiency of Liver, kidney, heart, lung, and brain function;
7. Patients with Severe anemia, dehydration, and severe disturbance of nutrient metabolism, which cannot be corrected or improved in the short term;
8. Patients with severe systemic infection, high fever (>38.5℃);
9. Pregnant and lactating women and those planning to become pregnant within one year;
10. Participants in clinical trials of any drugs and/or medical devices within 3 months before enrollment;
11. Any other factors that the investigator considers inappropriate for inclusion or that may affect the subject's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Ablation success rate | 1 month after ablation
  Ablation success rate = (numbers of nodule be completely ablated) / (numbers of nodule be ablated). Contrast-enhanced CT examination showed no significant enhancement of the nodule ablation area, and the nodule was considered to be completely ablated.

SECONDARY OUTCOMES:
Nodule ablation time | Immediately after ablation
  The time taken for nodule ablation is recorded according to the time displayed by the ablation instrument
Complete ablation rate | 3 months after ablation
  Ablation success rate = (numbers of nodule be completely ablated) / (numbers of nodule be ablated). Contrast-enhanced CT examination showed no significant enhancement of the nodule ablation area, and the nodule was considered to be completely ablated
Nodule recurrence rate | 6 months after ablation
  Ablation recurrence rate = (numbers of nodule recurrence) / (numbers of nodule be ablated). Contrast-enhanced CT showed the presence of an enhancement foci within the area of nodule ablation, and the nodule was considered to be recurrence.
Adverse events | Up to 6 months
  Adverse Events as assessed by NCI CTCAE V5.0 (Safety and Tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiao Liu, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No